CLINICAL TRIAL: NCT05889819
Title: Orange Almond Potato Cookies Supplementation Effect on the Height-for-Age Z-score Among Stunted Preschool-aged Children During COVID-19 Pandemic
Brief Title: Orange Almond Potato Cookies Supplementation
Acronym: CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Fatmah Fatmah, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaUniversity
Record Dates: First submitted 2023-05-13; First posted 2023-06-05 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Nutritional Stunting
Keywords: COVID19; stunted under-five children; weight; HAZ score; orange almond potato cookies
MeSH Terms: conditions — COVID-19; Body Weight

STUDY DESIGN:
Intervention Model Description: One treatment group received almond orange potato cookies during 4 weeks. One control group received almond potato cookies during 4 weeks.
Who Masked: Participant
Masking Description: Participants at the treatment and control groups received cookies supplementation during 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Intervention group received almond orange potato cookies during 4 weeks.
  Interventions: Dietary Supplement: Almond orange potato cookies for stunted under-five children
- Control group (Placebo Comparator): Control group received orange potato cookies during 4 weeks.
  Interventions: Dietary Supplement: Almond orange potato cookies for stunted under-five children

INTERVENTIONS:
Dietary Supplement: Almond orange potato cookies for stunted under-five children — Trained enumerator distributed 50 g cookies three times a week during 30 days to the treatment group.
  Anthropometry measurement: weight and height measured at pre study, during study (once a week), and post study.

SUMMARY:
The goal of this clinical trial is to assess the effect of potato almond orange cookie supplementation on the nutritional status of stunted under-five children.

The main questions aimed to answer are:

* Can cookie supplementation improve the weight of stunted under-five children?
* Can cookie supplementation improve the weight for age z score of stunted under-five children?

Participants divided in the two groups i.e.:

* Treatment group received 50 g potato almond orange cookie each day during 4 weeks.
* Control group received 50 g potato orange cookie each day during 4 weeks.
* Mothers of both groups given balanced nutrition education for stunted under-five children twice at the second and third week of study.

DETAILED DESCRIPTION:
Treatment group received 50 g potato almond orange cookie each day during 4 weeks.

Control group received 50 g potato orange cookie each day during 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age in the range of 12-59 months
* Male and female
* Lived in Sawangan Lama, Depok, and Depok Jaya neighborhoods of Depok City (three urban villages with a large stunting prevalence)
* Had a Height-for-Age Z-score (HAZ) index of < -2 SD
* Were not suffering from chronic or infectious diseases.

Exclusion Criteria:

* Suffered from chronic or infectious diseases

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Mean change of weight | 4 weeks
  Mean change of weight was measured by digital weighing SECA.
Mean change of height | 4 weeks
  Height was measured by microtoise.
Mean change of Height for Age - Z score | 4 weeks
  Height for Age - Z score was counted by WHO Anthro aplication

SECONDARY OUTCOMES:
Balanced nutrition of stunted under-five children knowledge | 4 weeks
  Mean change of mothers' knowledge on the balanced nutrition education measured by end-line questionnaire at the fourth week of study.

CONTACTS AND LOCATIONS:
Overall Officials: Fatmah Fatmah, Dr, Principal Investigator — Indonesia University
Locations (1):
- Depok, Depok Jaya, Sawangan Sub-districts, Depok, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No